CLINICAL TRIAL: NCT03478319
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of ACE-2494 in Healthy Postmenopausal Women
Brief Title: A Study of ACE-2494 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: A2494-01
Record Dates: First submitted 2018-03-07; First posted 2018-03-27 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: ACE-2494

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): ACE-2494 or placebo 0.06 mg/kg SC Day 1
  Interventions: Drug: ACE-2494 or placebo
- Cohort 2 (Experimental): ACE-2494 or placebo 0.2 mg/kg SC Day 1
  Interventions: Drug: ACE-2494 or placebo
- Cohort 3 (Experimental): ACE-2494 or placebo 0.6 mg/kg SC Day 1
  Interventions: Drug: ACE-2494 or placebo
- Cohort 4 (Experimental): ACE-2494 or placebo 1.0 mg/kg SC Day 1
  Interventions: Drug: ACE-2494 or placebo
- Cohort 5 (Experimental): ACE-2494 or placebo 2.0 mg/kg SC Day 1
  Interventions: Drug: ACE-2494 or placebo
- Cohort 6 (Experimental): ACE-2494 or placebo TBD (not to exceed 3.0 mg/kg SC) Day 1
  Interventions: Drug: ACE-2494 or placebo

INTERVENTIONS:
Drug: ACE-2494 or placebo — Recombination fusion protein

SUMMARY:
The purpose of the study is to assess safety, tolerance, pharmacokinetic, and pharmacodynamics of single doses of ACE-2494 in healthy postmenopausal women.

DETAILED DESCRIPTION:
Subjects will be evaluated for study inclusion/exclusion criteria during the screening period (within 4 weeks prior to Day -1) and eligible subjects who have signed the informed consent form (ICF) will be enrolled and treated with study drug (ACE-2494 or placebo) on Day 1. Subjects will be randomized (3:1, ACE-2494: placebo) to receive one dose of either ACE-2494 or placebo, respectively, on Day 1.

The primary objective of the study is to evaluate the safety and tolerability of single ascending doses of ACE-2494 in healthy postmenopausal women. The secondary objectives are to characterize the pharmacokinetic (PK) profile and pharmacodynamic (PD) effects, including serum biomarkers, fat, lean, and bone mass (DXA), muscle volume and intramuscular fat fraction (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women, with menopause defined by follicle stimulating hormone (FSH) level > 40 IU/L and either 12 months of spontaneous amenorrhea or at least 6 months post-surgical bilateral oophorectomy and/or hysterectomy
2. Age 45-75 years
3. Body mass index (BMI) 18.5-32.0 kg/m2
4. Clinical laboratory values that meet the following criteria prior to dosing on Day 1:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2 x upper limit of normal (ULN)
   2. Serum creatinine ≤ 1.5 x ULN
5. Ability to adhere to the study visit schedule/procedures, and to understand and comply with protocol requirements
6. Signed written informed consent

Exclusion Criteria:

1. Smokers (use of tobacco products within 3 months prior to screening)
2. History of hepatitis B (HBsAg and HB core Ab), human immunodeficiency virus (HIV) antibody or active hepatitis C
3. Positive drug or alcohol screen test at screening or on Day 1
4. History of drug or alcohol abuse (as defined by the investigator) or required treatment for drug or alcohol use within 2 years of Day 1
5. Donated or lost ≥ 500 mL of whole blood within 2 months prior to Day 1
6. History of opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia) within 6 months prior to screening; serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening
7. History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or any other drugs
8. Systemic glucocorticoid therapy, statin medication, growth hormone, androgen, insulin, oral hormone replacement therapy or any other therapy (including investigational) with known or intended effects on muscle within 3 months prior to Day 1
9. Anti platelet, anti-coagulant, or any other therapy (including investigational) with known or intended effects on bleeding risk within 1 week prior to Day 1 (Daily low-dose aspirin is allowed)
10. Treatment with another investigational drug, device, or approved therapy for investigational use within 30 days prior to Day 1; administration of a biological product in the context of a clinical research study within 90 days prior to Day 1
11. Participation in another clinical trial involving intervention with or without an investigational drug or device at any time during the study period
12. Unwilling or unable to maintain physical activity at baseline level for the duration of the study
13. For Cohorts 4-6 only, any condition that would prevent MRI scanning or compromise the ability to obtain a clear and interpretable scan of the thigh (e.g., pacemaker, knee/hip replacement, metallic implant, extreme claustrophobia, etc.)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with ACE-2494 treatment-related adverse events as assessed by CTCAE v5.0 | From initiation of treatment (Study Day 1) to end of follow-up period (Study Day 85)
  Adverse events (including both clinical observations and laboratory measurements), deemed related to ACE-2494 treat, will be recorded for each study subject

SECONDARY OUTCOMES:
Determination of ACE-2494 serum Cmax | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Determination of maximum serum concentration of ACE-2494 following subcutaneous administration
Determination of ACE-2494 serum Tmax | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Determination of time to maximum serum concentration of ACE-2494 following subcutaneous administration
Determination of ACE-2494 serum T1/2 | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Determination of serum half-life of ACE-2494 following subcutaneous administration
Determination of ACE-2494 AUC | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Determination of the area under the serum concentration curve of ACE-2494 following subcutaneous administration
Quantitation of serum GDF8 following ACE-2494 treatment | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Quantitation of serum levels of growth differentiation factor (GDF)8 following treatment with ACE-2492
Quantitation of serum BSAP following ACE-2494 treatment | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Quantitation of serum levels of bone-specific alkaline phosphatase (BSAP) following treatment with ACE-2494
Quantitation of serum CTX following ACE-2494 treatment | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Quantitation of serum levels of carboxy-terminal collagen crosslinks (CTX) following treatment with ACE-2494
Quantitation of serum FSH following ACE-2494 treatment | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Quantitation of serum levels of follicle stimulating hormone (FSH) following treatment with ACE-2494
Determination of body composition following ACE-2494 treatment by DXA | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Regional and whole-body quantitation of fat mass by dual energy X-ray absorptiometry (DXA) following treatment with ACE-2494
Determination of body composition following ACE-2494 treatment by DXA | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Regional and whole-body quantitation of lean mass by dual energy X-ray absorptiometry (DXA) following treatment with ACE-2494
Determination of body composition following ACE-2494 treatment by DXA | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Regional and whole-body quantitation of bone mass by dual energy X-ray absorptiometry (DXA) following treatment with ACE-2494
Determination of thigh muscle volume and intramuscular fat following ACE-2494 treatment by MRI for patients in Cohorts 4-6 only | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Determination of total muscle volume in the thigh by magnetic resonance imaging (MRI)
Determination of thigh muscle volume and intramuscular fat following ACE-2494 treatment by MRI for patients in Cohorts 4-6 only | From initiation of treatment, Study Day (SD)1 to end of follow-up period (SD85)
  Determination of intramuscular fat in the thigh by magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Québec, Canada